CLINICAL TRIAL: NCT01423266
Title: Examining the Effects of a High Protein Diet on Adiposity and Cardiac Structure in Patients With Heart Failure, Obesity, and Diabetes Mellitus
Brief Title: Effects of a High Protein Diet on Clinical Outcomes in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lorraine Evangelista, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01HL093466-01 (NIH)
Record Dates: First submitted 2011-08-15; First posted 2011-08-25 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Heart Failure; Diabetes Mellitus
Keywords: High Protein Diet in heart failure; obesity and heart failure; Weight management in Heart failure; heart failure, diabetes and obesity
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Protein Group (Experimental): 12-week supervised weight loss program consisting of a HP diet defined as 30% of energy from protein, 40% from carbohydrates and 30% from fat
  Interventions: Procedure: 12-week supervised weight loss intervention
- Standard Protein Group (Active Comparator): 12-week supervised weight loss program consisting of a SP diet defined as 15% of energy from protein, 55% from carbohydrates and 30% from fat
  Interventions: Procedure: 12-week supervised weight loss intervention

INTERVENTIONS:
Procedure: 12-week supervised weight loss intervention — Patients in the 2 study arms will participate in an intensive 12-week supervised weight loss intervention and will be seen by the same dietician at regular intervals: baseline, 2 weeks, 4 weeks, 8 weeks, and 12 weeks. Participants will receive personalized nutrition counseling and support during each of these visits. Participants will be randomized to either the HP or SP diet and assigned to receive one of two standard structured energy-restricted meal plans (1200, 1500 Kcal/day) based on the computed calorie deficit
  Other Names: weight management; diet; nutritional supervision

SUMMARY:
This research project was designed to study the role of dietary modifications in heart failure (HF) patients that suffer from type 2 diabetes mellitus and obesity. Specifically, the purpose of this study is to determine whether or not heart failure patients participating in a 3-month intensive lifestyle modification program of either a high protein (30 % of total calories from protein) group will have a significant improvement in weight reduction, quality of life and clinical outcomes compared to a standardized protein (15% of total calories from protein) group.

DETAILED DESCRIPTION:
Clinical management of heart failure (HF) related to obesity and diet recommendations currently lacks a strong scientific basis, and clinicians are divided in their approach to diet recommendations for this patient population. It has been shown that in extremely obese HF patients, weight reduction improves cardiac structure and function as well as functional status and symptomatology. Evidence on the impact of voluntary weight loss on improvement in survival in obese HF patients, however, is limited.

The purpose of this study is to determine whether or not heart failure patients participating in a 3-month intensive lifestyle modification program of either a high protein (30% of total calories from protein) group will have a significant improvement in weight reduction, quality of life and clinical outcomes compared to a standardized protein (15% of total calories from protein) group.

In addition to dietary interventions, participants in both groups with be given an exercise prescription and encouraged to exercise for 20-30 minutes at least 3-5 times each week as tolerated. They will also continue to receive usual medical care, advice and other support for their condition from their cardiologist or medical physician. Both sets of participants will utilize self-monitoring tools to assist with diet compliance and behavior change. These self-monitoring tools are mandatory and will be collected and analyzed. At each visit, subjects will also be asked to will also be asked to have their weight and waist circumference measured and, at select visits, they will provide a 24 hour recall to assess fullness with the overall diet. Subjects will be given a 3-day food (3DFR) record at baseline, which will be returned at the the 2-week, 4- week and 8-week visits, and will also complete the 3DFR at three months.

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI > 27 kg/m2);
* history of type 2 DM or documented impaired fasting glucose (IFG) according to fasting plasma glucose levels of 100-125 mg/dl or meeting 3 out of 4 criteria or Metabolic Syndrome ( as defined by the International Diabetes Federation 2011
* evaluation of HF and optimization of medical therapy; and
* ischemic or idiopathic HF etiology.

Exclusion Criteria:

* age ≤18 years old;
* history of clinically significant illness including acute myocardial infarction or sustained ventricular arrhythmia in the prior 3 months or current liver, respiratory, and/or gastrointestinal disease and malignancy;
* pregnancy or lactation;
* serum creatinine level > 1.5 mg/dl;*
* currently participating in a supervised weight loss program;
* physician refusal to permit patient participation in the study; and
* weight loss of >6% in the last 6 months
* gout or history of gout

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in adiposity (and body composition; i.e., % body fat)) | 3 months and 15 months

SECONDARY OUTCOMES:
Change from Baseline in lipid profiles (while controlling for statin drug dosage) | 3 months and 15 months
Change from Baseline in glycemic control and insulin resistance | 3 months and 15 months
Change from Baseline in peripheral blood circulation (as measured using peripheral arterial tonometry and plasma nitroxide measurement) | 3 months and 15 months
Change from Baseline in levels of quality of life | 3 months and 15 months

OTHER OUTCOMES:
Change in Cardiac Structure | 3 months and 15 months
Change in Cardiac Function | 3 months and 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine S Evangelista, PhD,RN,FAAN, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data management and analysis is in progress.